CLINICAL TRIAL: NCT02051010
Title: ABC Survey: Are we Meeting the Needs of Patients With Advanced Breast Cancer (ABC) in Ireland? A Nationwide Survey
Brief Title: ABC Survey - do we Meet the Needs of Patients With Advanced Breast Cancer?
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 13-01
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic Breast Cancer

SUMMARY:
The study will follow a descriptive design involving a survey. Data collection will involve paper based questionnaires. The questionnaires have been developed in conjunction with breast cancer support groups associated with the Irish Cancer Society and patients.

DETAILED DESCRIPTION:
The purpose of the study is to identify and categorise the need of Metastatic Breast Cancer (MBC) patients in Ireland with particular focus on; quality of life, symptom burden and access to and value of support available.

The study also aims to evaluate future service developments that will provide support to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Clinical diagnosis of MBC
* Female aged 18 years or older
* Able to complete the questionnaires independently

Exclusion Criteria:

* Any patient who does not meet the above mentioned inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients must have metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Needs of MBC patients in Ireland | Following analysis of the questionnaires completed by the patients, estimated 24 months
  The needs of MBC patients to be identified and categorised with particular focus on; quality of life, symptom burden and access to and value of available support

SECONDARY OUTCOMES:
Future service developments | Following analysis of the questionnaires completed by patients, estimated 24 months
  Evaluation of future service developments that will provide support to these patients

CONTACTS AND LOCATIONS:
Locations (13):
- Ireland (13):
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - South Infirmary - Victoria University Hospital, Cork
  - Letterkenny General Hospital, Donegal
  - Saint Vincent Universtiy Hospital, Dublin
  - Mater Misericordiae University Hospital and Mater Private Hospital, Dublin
  - Saint James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Galway University Hospital, Galway
  - Kerry General Hospital, Kerry
  - Midwestern Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford